CLINICAL TRIAL: NCT00438646
Title: Oral Bacteria and History of Allergic Disease in Children: A Pilot Study
Brief Title: Oral Bacteria and Allergic Disease in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907109; 07-E-N109
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2008-11

CONDITIONS: Asthma; Rhinitis; Eczema; Respiratory Sounds; Hypersensitivity
Keywords: Allergy; Asthma; Eczema; Hay Fever; Epidemiology
MeSH Terms: conditions — Asthma; Rhinitis; Eczema; Respiratory Sounds; Hypersensitivity; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will see if bacteria differ between children who have allergies or asthma and children who do not have allergies or asthma. Previous research suggests that some bacteria may protect against allergies and asthma. This study may provide more information on why some children develop allergies and asthma.

Patients at the University of North Carolina-Chapel Hill School of Dentistry who are between 6 and 11 years of age may be eligible for this study.

Parents of participating children complete a questionnaire about the child and the child's health. The child provides a saliva sample by chewing a small piece of wax and spitting in a cup.

The saliva sample is analyzed in the laboratory for bacteria, yeast and antibodies (substances the body produces to fight germs).

...

DETAILED DESCRIPTION:
The purpose of this study is to examine the feasibility of and to establish methods for a future study that will investigate associations between oral bacteria and allergic diseases in children. Rates of allergic diseases such as asthma, hay fever, and eczema have increased in the U.S. over the past several decades. One explanation for those increases is the Hygiene Hypothesis, which contends that decreases in microbial exposures have made the population more reactive to environmental allergens. Reports of protective associations for various infections and exposures to farms, pets, siblings, and day care have provided support for the Hypothesis. Preliminary work by NIEHS researchers suggests that some oral bacterial exposures may be beneficial. NIEHS researchers recently reported that elevated serum antibody concentrations to two common oral pathogens were associated with lower prevalences of asthma, wheeze, and hay fever in the U.S. population. Using a mouse model, NIEHS researchers found that immune responses involved in allergic airway inflammation could be modulated by infection with an oral pathogen. To further investigate these associations in humans, NIEHS researchers, in collaboration with UNC researchers, are planning an observational study that will collect saliva samples from and allergy information on child patients at the UNC-Chapel Hill School of Dentistry. Because we anticipate that several hundred children might have to be enrolled, we are proposing to test methods in a pilot study of 60 children. Twenty children will be recruited from each of three pediatric clinics. A research assistant will obtain the parent's consent and the child's assent and administer a questionnaire to the parent. The child's dentist will collect one teaspoon of saliva by having the child chew a piece of inert wax and spit into a sterile collection cup. Samples will be transported to the NIEHS and analyzed for bacterial species and for allergy-related cytokines. The specific aims for this pilot study are: 1) to identify the most efficient recruitment strategies, 2) to estimate response rates, 3) to estimate the distribution of allergic diseases among the children, 4) to identify any problematic consent form and questionnaire items, 5) to optimize saliva collection and laboratory protocols, and 6) to estimate statistical parameters required for more precise sample size calculations. Information gained from this pilot study will allow us to decide whether a larger study among this clinic population is feasible and to design a more efficient study if we decide to proceed.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Aged 6-11 years.
  2. Child is presenting to the UNC-CH School of Dentistry for a scheduled appointment.
  3. Sibling has not been enrolled.
  4. Parent consents to child's participation.
  5. Parent is willing to provide answers to a questionnaire.
  6. Child assents to the study.
  7. Child is willing and able to provide a usable saliva sample.

EXCLUSION CRITERIA:

1. Child is unwilling or unable to provide a usable saliva sample.
2. Parent or child is non-English speaking.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2007-02; Primary Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Mannino DM, Homa DM, Akinbami LJ, Moorman JE, Gwynn C, Redd SC. Surveillance for asthma--United States, 1980-1999. MMWR Surveill Summ. 2002 Mar 29;51(1):1-13. PMID 12420904
- [Background] Arbes SJ Jr, Gergen PJ, Elliott L, Zeldin DC. Prevalences of positive skin test responses to 10 common allergens in the US population: results from the third National Health and Nutrition Examination Survey. J Allergy Clin Immunol. 2005 Aug;116(2):377-83. doi: 10.1016/j.jaci.2005.05.017. PMID 16083793
- [Background] Liu AH, Murphy JR. Hygiene hypothesis: fact or fiction? J Allergy Clin Immunol. 2003 Mar;111(3):471-8. doi: 10.1067/mai.2003.172. PMID 12642824